CLINICAL TRIAL: NCT00819468
Title: Pharmacokinetics of 20 mg Teduglutide in Subjects With Moderately Impaired Hepatic Function Compared to Healthy Subjects With Normal Hepatic Function
Brief Title: Pharmacokinetics (PK) of 20 mg Teduglutide in Participants With Moderately Impaired Hepatic Function Compared to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CL0600-017
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — teduglutide; ALX-0600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participants with Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment (Child-Pugh score of 7-9) will receive 20 mg of teduglutide.
  Interventions: Drug: Teduglutide
- Healthy Volunteers (Active Comparator): Healthy volunteers with normal hepatic function matched to hepatic impaired participants by age, gender, BMI, and renal function as measured by creatinine will receive 20 mg of teduglutide.
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — Participants will receive 20 mg dose of lypholized powder of teduglutide mixed with sterile water and injected subcutaneously into the abdomen.
  Other Names: GATTEX

SUMMARY:
This is a study to compare the pharmacokinetic profile of teduglutide in healthy participants with normal hepatic function with participants who have moderate hepatic impairment.

DETAILED DESCRIPTION:
24 participants (equally divided between participants with normal hepatic function and those with moderate hepatic impairment (defined by the protocol as a Child-Pugh classification of grade B score of 7-9)will be given a single injection of teduglutide (20mg) through subcutaneous injection into the abdomen. Blood samples would be taken within 30 minutes of dose through 24 hours post-dose. Participants in both groups are matched up by sex, age, BMI, and renal function.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between 18 and 85 years of age
* BMI of 18 to 40, inclusive
* Creatinine clearance (greater) > 50 milliliter per minute(mL/min)
* Able to understand and willing to sign an informed consent form (ICF)
* Willing and able to be confined at the study site for approximately 2.5 days
* Female participants who are postmenopausal, surgically sterilized, or women of childbearing potential (WOCBP) using an effective form of birth control during the study
* WOCBP must have a negative urine beta human chorionic gonadotropin (β-hCG) result at screening (Days -28 to -2) and check-in (Day -1)
* Negative urine test for selected drugs of abuse and alcohol at screening and check-in (Day-1)

Inclusion for participants with Impaired Hepatic Function (in addition to above criteria):

* Documented moderately impaired hepatic function defined by a total score of 7 to 9 on the Child-Pugh Classification at screening and check-in
* No clinically significant change in disease status within the 3 months prior to study entry
* Abnormal laboratory results that are related to the participants underlying condition clinically stable as deemed by the investigator
* Abstained from alcohol use within 90 days prior to study entry when hepatic impairment is known to be secondary to alcohol abuse
* On medication and/or treatment regimen if, in the opinion of the investigator, the underlying disease is under control
* Participants with normal hepatic function will be matched collectively as a group by gender, age, and BMI with the participants with moderately impaired hepatic function. Participants with normal hepatic function will also be matched on an individually with the participants with moderately impaired hepatic function with regard to renal function In addition to inclusion criteria # 1 to 8, participants with normal hepatic function must also meet the following inclusion criteria to be eligible for participation in this study:
* Similar level of renal function based on Cockroft-Gault equation as the matched participant with moderately impaired hepatic function
* Medically healthy with normal or clinically insignificant clinical results at screening and check-in

Exclusion Criteria:

* Donated 1 pint or more of blood or blood products within 7 days prior to the study, and/or had a blood or plasma donation within 7 days prior to the study
* Participated in any other investigational drug trial within 30 days prior to study entry
* Have a hemoglobin level < 10.0 g/dL at screening (Days -28 to -2)
* Have any condition that, in the opinion of the investigator or sponsor, would make them unsuitable for the study
* Participants with Impaired Hepatic Function (in addition to exclusion criteria 1-4):
* Acceptable Child-Pugh score (Grade B, score of 7 to 9), which is associated with conditions such as metastatic cancer rather than impaired hepatic function
* Participants with Normal Hepatic Function (in addition to exclusion criteria 1-4
* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* History or evidence of congenital nonhemolytic hyperbilirubinemia
* History or evidence of gallstone disease or stomach or intestinal surgery, with the exception of appendectomy
* History or evidence of colorectal cancer
* History or evidence of malabsorption, pancreatic disease or gastrointestinal disorders, such as irritable bowel syndrome, Crohn's disease or ulcerative colitis
* Taking prescription or over-the-counter medication (with the exception of daily low dose aspirin regimen and/or birth control)during the 7 days preceding confinement to the clinical research unit, and/or who anticipate a need to use prescription or over-the-counter medication during the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-07-26 (Actual); Primary Completion 2007-08-23 (Actual); Study Completion 2007-08-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve From Time Zero to Time of the Last Measurable Concentration (AUC0-last) | Pre-dose, 3 hours and 24 hours post-dose
  AUC0-last of Teduglutide will be evaluated.
Maximum concentration (Cmax) | Pre-dose, 3 hours and 24 hours post-dose
  Cmax of Teduglutide will be evaluated.
Elimination Half-Life (t1/2) | Pre-dose, 3 hours and 24 hours post-dose
  t1/2 of Teduglutide will be evaluated.

SECONDARY OUTCOMES:
Number of participants with Adverse events (AEs) | From start of study treatment to follow up (up to 9 days)
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical/medicinal product which includes an exacerbation of a pre-existing illness, sign, symptom, or clinically significant laboratory test abnormality that is detected or diagnosed after study drug administration, pretreatment or post-treatment events that occur as a result of protocol-mandated procedures. An AE does not necessarily have to have a causal relationship with study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- University of Miami Clinical Pharmacology Unit, Miami, Florida, United States